CLINICAL TRIAL: NCT07101380
Title: A Multicenter, Prospective, Investigator-initiated, Feasibility Randomized Controlled Study to Evaluate the Applicability and Safety of the Multi-Domain Personalized Physical Activity Prescription Software 'SuperBrain BOOM' for Patients With Mild Cognitive Impairment
Brief Title: Feasibility Study of 'SuperBrain BOOM' for Mild Cognitive Impairment Patients
Acronym: SuperBrainBOOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, So Young Moon, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AJOUIRB-DE-2025-36; RS-2024-00337993 (Other Grant/Funding Number: Korea Health Industry Development Institute)
Record Dates: First submitted 2025-07-25; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment; MCI; Physical Activity; SuperBrain BOOM; Digital Health; Dementia Prevention
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tablet-based intervention group (Experimental)
  Interventions: Device: Tablet-based Physical SuperBrain BOOM
- Smartphone-based intervention group (Experimental)
  Interventions: Device: Smartphone-based SuperBrain BOOM
- Control group (No Intervention)

INTERVENTIONS:
Device: Tablet-based Physical SuperBrain BOOM — This intervention is a tablet-based physical activity program designed for patients with Mild Cognitive Impairment (MCI).
  Participants receive a personalized exercise plan through a tablet application, with real-time feedback to enhance cognitive function.
  Compared to the smartphone-based version, this program is designed to provide a larger interface and structured environment, allowing participants to engage in the program using a tablet at home or in a clinical setting.
  The app also helps track progress and encourage adherence to the exercise regimen.
  Arms: Tablet-based intervention group
Device: Smartphone-based SuperBrain BOOM — This intervention is a smartphone-based physical activity program designed for MCI patients. Participants receive a personalized exercise plan through a smartphone app, with real-time feedback to enhance cognitive function. Unlike the tablet-based intervention, this program is designed to be more portable and flexible, enabling participants to engage in the program from anywhere using their smartphones. The app also helps track progress and encourage adherence to the exercise regimen.
  Arms: Smartphone-based intervention group

SUMMARY:
The goal of this clinical trial is to learn whether a mobile-based personalized physical activity program called SuperBrain BOOM is safe and works to improve cognitive function, physical performance, mood, and quality of life in older adults (ages 50-85) with mild cognitive impairment (MCI).

The main questions it aims to answer are:

Can SuperBrain BOOM be safely and effectively used by people with MCI? Does the program help improve cognitive and physical function? Do participants stay engaged and complete the program as expected?

Researchers will compare:

A mobile intervention group using SuperBrain BOOM (on tablet or smartphone) A control group receiving usual care

Participants will:

Use a tablet or smartphone to follow a personalized physical activity program for 12 weeks Complete clinical assessments on cognition, physical ability, mood, and nutrition Be monitored for safety and program adherence using automatically collected data

DETAILED DESCRIPTION:
This study is designed to assess the feasibility, safety, and potential benefits of a multi-domain personalized physical activity intervention-SuperBrain BOOM-delivered via mobile devices (tablet or smartphone) for individuals with Mild Cognitive Impairment (MCI).

Mild Cognitive Impairment is a condition in which individuals experience noticeable cognitive decline without significant impairment in daily functioning. It is considered a transitional stage between normal aging and dementia. Evidence suggests that regular physical activity and cognitive engagement can delay or reduce the risk of progression to dementia.

SuperBrain BOOM provides personalized exercise programs tailored to each participant's cognitive status, physical capacity, and lifestyle, and is designed to improve cognitive function, physical performance, emotional well-being, and quality of life.

This randomized controlled trial will allocate participants into three groups: a mobile intervention group (tablet or smartphone) and a control group receiving usual care. The primary outcomes include changes in cognitive function, physical performance, mood, nutritional status, and quality of life over 12 weeks. Safety and adherence will be monitored throughout the intervention using system-generated data and clinical assessments.

Secondary analyses will explore subgroup differences based on APOE genotype and demographic variables to better understand who benefits most from the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Between 50 and 85 years old.
2. Meets all of the core clinical criteria for suspected Mild Cognitive Impairment (MCI) according to the National Institute on Aging-Alzheimer's Association (NIA-AA) guidelines as of the screening date:

   * Concerns of the participant or caregiver regarding cognitive decline compared to prior functioning.
   * Impairment in at least one cognitive domain.
   * Preserved independence in overall daily living activities.
   * No dementia.
3. Has one or more of the following neuropsychological test results within one year of the screening date, with delayed recall scores in the memory domain below the mean -1.0 standard deviation according to age- and education-adjusted normative data:

   * Seoul Neuropsychological Screening Battery 2nd Edition (SNSB-II)
   * Korean version of the Consortium to Establish a Registry for Alzheimer's Disease (CERAD-K)
   * Literacy Independent Cognitive Assessment (LICA)
4. As of the screening date, has a Korea-Mini Mental State Examination (K-MMSE-2) score that corresponds to at least -1.5 standard deviations below the mean based on age- and education-adjusted normative data.
5. As of the screening date, has a Global Clinical Dementia Rating (CDR) score of 0.5, with a memory score of either 0.5 or 1.
6. Capable of using a tablet or smartphone with training, or has a research partner who can assist with using a tablet or smartphone.
7. Has a caregiver who regularly contacts the participant:

   -A caregiver who is able to support the participant (monitor compliance and report participant status) and spends at least 8 hours per week with the participant during the trial period.
8. The participant provides written informed consent to participate in the study.

Exclusion Criteria:

1. Presence of psychiatric disorders, such as major depression.
2. Dementia.
3. Other neurodegenerative diseases, such as Parkinson's disease.
4. Malignant tumors within the past 5 years that have not been declared cured.
5. Vascular surgery or stent placement within the past year.
6. Severe or unstable symptomatic cardiovascular disease.
7. Evidence of severe or unstable physical conditions, such as acute or severe asthma, active peptic ulcers, severe liver disease, kidney disease requiring dialysis, or any other medical conditions that may interfere with completing the clinical trial.
8. Severe vision impairment, severe hearing loss, or communication difficulties that would prevent the participant from undergoing the intervention or efficacy assessments.
9. Abnormal findings in clinical pathology tests related to cognitive decline, as determined by the clinical investigator (e.g., significant thyroid dysfunction, vitamin B12 or folate deficiency, neurosyphilis, etc.).
10. The investigator's judgment that the participant is unlikely to cooperate fully with the study.
11. The investigator's judgment that the participant has difficulty safely participating in an exercise-based intervention program.
12. Participation in another interventional clinical trial.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
14-item cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAS-cog14) | Baseline (Week 0, pre-intervention) and Week 12 (end of intervention)
  The ADAS-cog14 is a comprehensive cognitive assessment tool that includes memory, attention and concentration, planning and executive function, visuoconstruction, and orientation. Scores range from 0 to 90, with higher scores indicating worse cognitive function. The assessment will be conducted at baseline and at the end of the intervention (Week 12).

SECONDARY OUTCOMES:
Korean Mini-Mental State Examination, 2nd Edition (K-MMSE-2) | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  The Korean Mini-Mental State Examination, 2nd Edition (K-MMSE-2), is a brief cognitive screening tool widely used to assess general cognitive function. It evaluates orientation, memory, attention and calculation, visuospatial ability, and language through verbal and written tasks. Scores range from 0 to 30, with higher scores indicating better cognitive function. The assessment will be conducted at screening and at the end of the intervention (Week 12).
Clinical Dementia Rating scale - Sum of Boxes (CDR-SB) | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  The Clinical Dementia Rating scale - Sum of Boxes (CDR-SB) is used to assess the overall severity of dementia across six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The total score ranges from 0 to 18, with higher scores indicating more severe cognitive impairment. The assessment will be conducted at screening and at the end of the intervention (Week 12).
Korean Instrumental Activities of Daily Living (K-IADL) | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  The Korean Instrumental Activities of Daily Living (K-IADL) is an 11-item assessment tool used to evaluate functional independence in daily life activities, including telephone use, shopping, food preparation, housekeeping, and medication management. Each item is scored from 0 to 3, and a mean score of 0.4 or higher suggests possible dementia. Higher scores indicate greater impairment in instrumental activities of daily living. The assessment will be conducted at screening and at the end of the intervention (Week 12).
Timed Up and Go test | Baseline (Week 0, pre-intervention) and Week 12 (end of intervention)
  The Timed Up and Go (TUG) test is used to assess mobility and balance. Participants are seated on a chair placed 3 meters from a cone, with both feet on the ground and hands on their thighs. At the signal to start, they rise from the chair, walk to the cone, circle it, return, and sit down. After a demonstration and one practice trial, the test is performed twice, and the better of the two times (in 0.1-second units) is recorded. The assessment will be conducted at baseline and at the end of the intervention (Week 12).
30-second Sit-to-Stand Test | Baseline (Week 0, pre-intervention) and Week 12 (end of intervention)
  The 30-second sit-to-stand test is used to assess lower body strength and endurance. Participants sit in a chair with arms crossed over the chest and hands resting on the shoulders. They are instructed to fully stand up and sit down as many times as possible within 30 seconds, keeping the knees, hips, and back extended. The number of repetitions is automatically recorded by the app. The test will be conducted at baseline and at the end of the intervention (Week 12).
2-Minute Step Test | Baseline (Week 0, pre-intervention) and Week 12 (end of intervention)
  The 2-Minute Step Test is used to assess aerobic endurance. Participants are instructed to march in place for 2 minutes, lifting their knees to a height midway between the patella (kneecap) and iliac crest (hip). Each time the right knee reaches the required height, one count is recorded. The final score is calculated by dividing the total step count by 2. The test will be conducted at baseline and at the end of the intervention (Week 12).
Quality of Life-Alzheimer's Disease (QOL-AD) | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  The Quality of Life-Alzheimer's Disease (QOL-AD) scale is a 13-item questionnaire designed to assess the quality of life in individuals with Alzheimer's disease. It includes both self-report from the participant and proxy-report from a caregiver. Total scores range from 0 to 52, with higher scores indicating better perceived quality of life. The assessment will be conducted at screening and at the end of the intervention (Week 12).
Nutritional Quotient for Elderly (NQ-E) | Baseline (Week 0, pre-intervention) and Week 12 (end of intervention)
  The Nutritional Quotient for Elderly (NQ-E) is a 20-item self-administered questionnaire developed to comprehensively assess dietary quality and nutritional status in older adults. Participants are asked to read and respond to items related to dietary behaviors, balance, diversity, moderation, and dietary environment. The total score ranges from 0 to 100, with higher scores indicating better nutritional status and quality of diet. The assessment will be conducted at baseline and at the end of the intervention (Week 12).
Mini Nutritional Assessment (MNA) | Baseline (Week 0, pre-intervention) and Week 12 (end of intervention)
  The Mini Nutritional Assessment (MNA) is a validated screening tool for evaluating nutritional status in older adults. It includes questions on recent food intake, weight loss, mobility, psychological stress, and body mass index (BMI). The total score ranges from 0 to 14, with higher scores indicating better nutritional status. The assessment will be conducted at baseline and at the end of the intervention (Week 12).
Assessment of Metabolic and Vascular Risk Factors | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  This assessment includes vital signs and anthropometric measurements (blood pressure, waist circumference, weight, body mass index), as well as lifestyle factors (alcohol consumption and smoking status). Additionally, blood tests will be conducted to evaluate metabolic and vascular risk markers, including fasting glucose, HbA1c, total cholesterol, triglycerides, HDL-C, LDL-C, BUN, and creatinine. Blood samples (8 cc) will be collected at screening and at the end of the intervention and analyzed by Seoul Clinical Laboratories. Higher levels of glucose, lipids, or renal markers may indicate elevated cardiometabolic risk.
Geriatric Depression Scale-15 items (GDS-15) | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  The Geriatric Depression Scale-15 items (GDS-15) is a self-report screening tool designed to assess depressive symptoms in older adults. Participants respond "yes" or "no" to 15 questions related to mood, energy, and interest. Total scores range from 0 to 15, with higher scores indicating greater severity of depressive symptoms. In the Korean validation study, a score of 8 or higher suggests the possibility of depression. The assessment will be conducted at screening and at the end of the intervention (Week 12).
Prospective and Retrospective Memory Questionnaire (PRMQ) | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  The Prospective and Retrospective Memory Questionnaire (PRMQ) is a 16-item self- and proxy-report questionnaire that assesses everyday memory performance. Each item is rated on a 5-point scale (1 to 5), with total scores ranging from 16 to 80. Lower scores indicate better memory function, while higher scores suggest more frequent memory failures. Both the participant and a caregiver will complete the questionnaire at screening and at the end of the intervention (Week 12).
Pittsburgh Sleep Quality Index (PSQI) | Screening (within 14 days prior to baseline) and Week 12 (end of intervention)
  The Pittsburgh Sleep Quality Index (PSQI) is a 7-component self-report questionnaire used to assess subjective sleep quality over the past month. It evaluates sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored from 0 to 3, and the total score ranges from 0 to 21. A total score of 8 or less indicates good sleep quality, while a score of 9 or higher suggests poor sleep quality. The assessment will be conducted at screening and at the end of the intervention (Week 12).

CONTACTS AND LOCATIONS:
Overall Officials: So Young Moon, Principal Investigator — Ajou University School of Medicine
Locations (5):
- South Korea (5):
  - Bundang CHA General Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Kangwon National University Hospital, Chuncheon
  - Chonnam National University Hospital, Gwangju

IPD SHARING:
Plan to Share IPD: No